CLINICAL TRIAL: NCT05638139
Title: Treatment of Ano-perineal Fistulas Resistant to Surgical Treatment with a Gel and Plug of Wharton's Jelly
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TBF Genie Tissulaire (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SygeLIX-Fistules-TBF; 2021-A02787-34 (Other: IDRCB)
Record Dates: First submitted 2022-11-24; First posted 2022-12-06 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Anal Fistula
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SygeLIX-F + SygeLIX-G (Experimental): Combination of SygeLIX-F, a plug made of an assembly of umbilical cord lining and Wharton's jelly in the form of a cylinder of porous structure, and SygeLIX-G, a Wharton's jelly gel reconstituted in a syringe.
  Interventions: Biological: SygeLIX-F + SygeLIX-G

INTERVENTIONS:
Biological: SygeLIX-F + SygeLIX-G — SygeLIX-F (plug) is inserted through the internal orifice while cryptoglandular space is filled by SygeLIX-G (gel).

SUMMARY:
The purpose of this open, multicenter pilot trial is to evaluate the tolerance of the combination of a gel and a plug made of Wharton's jelly in the treatment of ano-perineal fistulas resistant to surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 to 65 years.
* Patient with a single anal fistula resistant after at least one surgical treatment. Fistula may be related to Crohn's disease.
* Patient with an upper transsphincteric or lower transsphincteric fistula.
* Patient presenting fistula with or without intersphincteric diverticula.
* Fistula effectively drained with a seton.
* Informed and consenting patient.
* Patient who is a member or a beneficiary of a national health insurance plan.

Exclusion Criteria:

* Pregnant or breastfeeding woman or woman of childbearing age without effective contraception.
* Patients who have had more than one failed obstruction technique.
* Patient with more than one internal orifice.
* Patient with an MRI proven abscess.
* Patient with an uncontrolled infection.
* Patient with a contraindication to anesthesia.
* Person deprived of liberty by a judicial or administrative decision.
* Adult subjected to a legal protection measure or unable to express his / her consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-06-27 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Evaluation of intensity of perineal inflammation following treatment | Through study completion (45 days)
  Scoring of pain (0 = no pain, 10 = worst pain possible), redness (0 = no redness, 4 = redness covering an area > 5 cm), edema (0 = no edema, 4 = area completely swollen), ulceration (0 = no ulceration, 4 = ulcer larger than 1 cm).
Rate of plug expulsion and surgical revision due to complications | Through study completion (45 days)
Type and incidence of adverse events (AE) and serious adverse events (SAE) | Through study completion (45 days)

SECONDARY OUTCOMES:
Evaluation of surgical technique | Time of investigational products surgical implantation (Day 0)
  Questionnaire on surgical technique including ease of plug suture to the mucosa and of gel use.
Plug integration | 30 days, 45 days
  Assessment of anal continence by the Vaizey score (0 = perfect continence, 24 = totally incontinent).
Cessation of fistula flow | 45 days
  Healing of the fistula orifices assessed by palpation and pinching.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Clinique Blomet, Paris
  - Maison de Santé Protestante de Bordeaux-Bagatelle, Talence

IPD SHARING:
Plan to Share IPD: No